CLINICAL TRIAL: NCT04293159
Title: Effect of Probiotic on Constipation and on Neuropsychological Performance in Patients With Parkinson's Disease
Brief Title: Effect of Probiotic on Constipation in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salerno (Other)
Collaborators: Roberto Erro (Unknown); Maria Teresa Pellecchia (Unknown); Antonella Santonicola (Unknown); Carolina Ciacci (Unknown)
Responsible Party: Principal Investigator, PAOLA IOVINO, Associate Professor, University of Salerno
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: University of Salerno
Record Dates: First submitted 2020-02-19; First posted 2020-03-03 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease; Constipation
Keywords: constipation; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Constipation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lactobacillus casei DG (Enterolactis duo®) (Experimental): Lactobacillus casei DG (Enterolactis duo®)
  Interventions: Dietary Supplement: Lactobacillus casei DG (Enterolactis duo®)

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei DG (Enterolactis duo®) — Lactobacillus casei DG (Enterolactis duo®)

SUMMARY:
The aim of the study is to collect data for the assessment of the Lactobacillus casei DG (Enterolactis ®duo) effect on constipation and on neuropsychological performance

DETAILED DESCRIPTION:
The aim of the study is to collect data for the assessment of the Lactobacillus casei DG (Enterolactis® duo) effect on overall abdominal pain, bowel movements and other abdominal symptoms and on neuropsychological performance in patients with Parkinson's Disease. The investigators suppose that, due to the immunomodulatory action of probiotics, overall neuropsychological function will improve as well as due also to prebiotic abdominal symptoms will decrease following consumption of Lactobacillus casei DG (Enterolactis® duo).

ELIGIBILITY:
Inclusion Criteria:

* A positive diagnosis of functional constipation or Irritable Bowel Syndrome -subtype constipation according to Rome IV criteria.
* Negative for colon cancer screening
* Negative relevant additional screening or consultation whenever appropriate.
* Ability of conforming to the study protocol.
* Stable treatment for Parkinson's disease

Exclusion Criteria:

* Presence of any other relevant organic, systemic or metabolic disease (particularly significant history of cardiac, renal, oncology, endocrinology, metabolic or hepatic disease), or abnormal laboratory values that will be deemed clinically significant on the basis of predefined values a part from Parkinson's disease
* Ascertained intestinal organic diseases, including ascertained celiac disease or inflammatory bowel diseases (Crohn's disease, ulcerative colitis, diverticular disease, infectious colitis, ischemic colitis, microscopic colitis).
* Previous major abdominal surgeries.
* Inability to conform with protocol.
* Recent history or suspicion of alcohol abuse or drug addiction.
* Previous participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
satisfaction with therapy | 12 weeks
  A "satisfaction with therapy" score (on a 7-point Likert scale: 1 = extremely dissatisfied, 2 = very dissatisfied, 3 = dissatisfied, 4 = partially satisfied, 5 = satisfied, 6 = very satisfied, 7 = extremely satisfied)
Improvement after treatment | 12 WEEKS
  "Improvement after treatment" was evaluated with a global rating-of-change scale (-7 to +7: -7 = extremely worsened, 0 = unchanged,
  +7 = extremely improved). "Improvement after treatment" was defined by an increase in the global rating-of-change scale of ≥2 points.
neuropsychological function | 12 weeks
  The Non-Motor Symptoms Scale (NMSS) is a 30-item rater-based scale that assesses a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The NMSS measures the severity and frequency of non-motor symptoms across nine dimensions. The scale can be used for patients at all stages of PD.The total NMSS score ranges from 0 to 360, the worst.

SECONDARY OUTCOMES:
the Unified Parkinson Disease Rating Scale (UPDRS, italian version) | 12 WEEKS
  the Unified Parkinson Disease Rating Scale (UPDRS, italian version). The UPDRS is a rating tool used to gauge the course of Parkinson's disease in patients. A score of 199 on the UPDRS scale represents the worst (total disability) with a score of zero representing (no disability); The Non-motor-symptoms scale (NMSS, italian version)
M-PAC SYM | 12 WEEKS
  M-PAC-SYM)5 The Patient Assessment of Constipation Symptoms (scoring from 0 = absent to 4 = very strong)

CONTACTS AND LOCATIONS:
Overall Officials: PAOLA IOVINO, MD, Principal Investigator — University of Salerno
Locations (1):
- Aou Sangiovanni E Ruggi D'Aragona, Salerno, Italy

REFERENCES:
- [Result] Erro R, Picillo M, Vitale C, Amboni M, Moccia M, Longo K, Cozzolino A, Giordano F, De Rosa A, De Michele G, Pellecchia MT, Barone P. Non-motor symptoms in early Parkinson's disease: a 2-year follow-up study on previously untreated patients. J Neurol Neurosurg Psychiatry. 2013 Jan;84(1):14-7. doi: 10.1136/jnnp-2012-303419. Epub 2012 Sep 19. PMID 22993448
- [Result] Fasano A, Visanji NP, Liu LW, Lang AE, Pfeiffer RF. Gastrointestinal dysfunction in Parkinson's disease. Lancet Neurol. 2015 Jun;14(6):625-39. doi: 10.1016/S1474-4422(15)00007-1. PMID 25987282
- [Result] Martinez-Martinez MI, Calabuig-Tolsa R, Cauli O. The effect of probiotics as a treatment for constipation in elderly people: A systematic review. Arch Gerontol Geriatr. 2017 Jul;71:142-149. doi: 10.1016/j.archger.2017.04.004. Epub 2017 Apr 14. PMID 28467916
- [Result] Bellini M, Usai-Satta P, Bove A, Bocchini R, Galeazzi F, Battaglia E, Alduini P, Buscarini E, Bassotti G; ChroCoDiTE Study Group, AIGO. Chronic constipation diagnosis and treatment evaluation: the "CHRO.CO.DI.T.E." study. BMC Gastroenterol. 2017 Jan 14;17(1):11. doi: 10.1186/s12876-016-0556-7. PMID 28088179
- [Result] Neri L, Iovino P; Laxative Inadequate Relief Survey (LIRS) Group. Bloating is associated with worse quality of life, treatment satisfaction, and treatment responsiveness among patients with constipation-predominant irritable bowel syndrome and functional constipation. Neurogastroenterol Motil. 2016 Apr;28(4):581-91. doi: 10.1111/nmo.12758. Epub 2016 Feb 12. PMID 26867677
- [Result] Cappello C, Tremolaterra F, Pascariello A, Ciacci C, Iovino P. A randomised clinical trial (RCT) of a symbiotic mixture in patients with irritable bowel syndrome (IBS): effects on symptoms, colonic transit and quality of life. Int J Colorectal Dis. 2013 Mar;28(3):349-58. doi: 10.1007/s00384-012-1552-1. Epub 2012 Aug 12. PMID 22885882